CLINICAL TRIAL: NCT02257554
Title: Comparing Patients' and Surgeons' Expectations of Lumbar Spine Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-287
Record Dates: First submitted 2014-09-30; First posted 2014-10-06 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Lumbar Spine Surgery
Keywords: expectations
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: education — Discussion of surgical expectations with patients

SUMMARY:
The goals of this study are to assess concordance between the patient-surgeon pair regarding expectations of lumbar spine surgery.

DETAILED DESCRIPTION:
Low back pain is a prevalent medical condition afflicting primarily older adults but affecting all age groups and due to acute and non-acute diagnoses. Multiple possible conservative therapies exist; however, their major drawback is that the time required to advance therapy is often prolonged and accompanied by persistent disability and psychological suffering. Thus, some patients seek surgery after exhausting other therapies and some patients seek surgery earlier in their course. For both groups, decisions to undergo surgery are based on personal circumstances, perspectives, and expectations of outcome. Prior studies have shown that patients typically have high expectations of orthopedic surgery. Although high aspirations can be motivating, they also may predispose to poor outcomes if they are unrealistic and cause patients to become discouraged with recuperation time and ignore recommended lifestyle changes that avert progression of disease. Expectations that are too low, conversely, also may predispose to poor outcomes if patients lack motivation to participate in rehabilitation and to follow postop precautions. In order to achieve maximum benefit from surgery, patients and surgeons need to share an understanding of what is possible, probable, and realistic, and to join together and work toward the same goals. The primary objective of this proposed cross-sectional study is to assess the concordance between patients and their surgeons regarding expectations of lumbar spine surgery. Patients scheduled for lumbar surgery will be dichotomized according to whether they have acute versus non-acute conditions. Several days before surgery patients will complete the validated Lumbar Spine Surgery Expectations Survey measuring their physical and psychological expectations. Also before surgery their surgeons will complete the surgeon's version of the same survey for each patient. The main outcome will be a comparison of the concordance within each patient-surgeon pair according to acute versus non-acute groups based on the concordance correlation coefficient. Multivariate regression analysis based on the GEE method will be used to assess covariates.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they are ≥ 18 years old, speak English, and are scheduled for non-trauma-related lumbar spine surgery.

Exclusion Criteria:

* Patients will be excluded if they have cognitive deficits and cannot provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for lumbar spine surgery and their surgeons
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2014-09; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of Lumbar Spine Surgery Expectations Survey scores for patients and their surgeons. | participants will be surveyed before surgery, an expected average of 5 days
  comparison of patients and surgeons responses

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Mancuso CA, Cammisa FP, Sama AA, Hughes AP, Ghomrawi HM, Girardi FP. Development and testing of an expectations survey for patients undergoing lumbar spine surgery. J Bone Joint Surg Am. 2013 Oct 2;95(19):1793-800. doi: 10.2106/JBJS.L.00338. PMID 24088972